CLINICAL TRIAL: NCT00489944
Title: A Phase II Pilot Trial of Sutent, Tamoxifen, and Cisplatin in Patients With High-Risk Ocular Melanoma
Brief Title: Sunitinib, Tamoxifen, and Cisplatin in Treating Patients With High-Risk Ocular Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Diego Pacific Oncology & Hematology Associates (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000551559; POHA-0604
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-07

CONDITIONS: Intraocular Melanoma
Keywords: ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; iris melanoma; epithelioid cell intraocular melanoma; stage IIB intraocular melanoma; stage IIIA intraocular melanoma; stage IIIB intraocular melanoma; stage IIIC intraocular melanoma; stage IV intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Cisplatin; Sunitinib; Tamoxifen; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: cisplatin
Drug: sunitinib malate
Drug: tamoxifen citrate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as tamoxifen and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sunitinib together with tamoxifen and cisplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving sunitinib together with tamoxifen and cisplatin works in treating patients with high-risk ocular melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of adjuvant sunitinib malate, tamoxifen citrate, and cisplatin on disease-free survival and overall survival of patients with high-risk ocular melanoma who have undergone primary therapy.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a pilot study.

Patients receive oral sunitinib malate once daily on days 1-21, oral tamoxifen citrate twice daily on days 1-7, and cisplatin IV on days 2 and 3. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 2 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ocular melanoma

  * High-risk disease, defined by any of the following:

    * Large choroidal tumors with a basal diameter ≥ 16 mm and/or tumor thickness ≥ 10 mm (T3)
    * Extrascleral extension (T4)
    * Ciliary body involvement
    * Epithelioid cell type only
* Have undergone appropriate primary treatment for ocular melanoma
* No measurable metastatic disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,200/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 50 mL/min
* AST and ALT ≤ 3 times upper limit of normal
* Pancreatic enzymes normal
* Thyroid function normal or stable on replacement therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Cardiac ejection fraction ≥ 50% by MUGA or ECHO
* No myocardial infarction within the past 6 months
* No congestive heart failure requiring medication
* No history of pulmonary disease requiring supplemental oxygen
* No dyspnea at rest
* No active infection
* No chronic underlying immunodeficiency disease
* No other serious illness that would preclude patient safety, in the opinion of the investigator
* No other cancer within the past 5 years except nonmelanoma skin cancer or cervical cancer
* No thromboembolic disease within the past 6 months

PRIOR CONCURRENT THERAPY:

* No prior sunitinib malate, tamoxifen citrate, or cisplatin
* No other concurrent chemotherapy, radiotherapy, or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-05; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. McClay, MD, Principal Investigator — San Diego Pacific Oncology & Hematology Associates
Locations (1):
- San Diego Pacific Oncology and Hematology Associates, Incorporated - Encinitas, Encinitas, California, United States